CLINICAL TRIAL: NCT00170482
Title: In Depth Immunologic Studies in Elderly Subjects Receiving Either Standard-Dose Fluzone (15mcg HA/Virus Strain) or High-Dose (60 mcg HA/Virus Strain) Trivalent Inactivated Influenza Virus Vaccine
Brief Title: Elderly Influenza Vaccine Immunogenicity Substudy
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 05-0028
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2011-04-26

CONDITIONS: Influenza
Keywords: Fluzone; inactivated; influenza vaccine; sub-study; trivalent
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Time Perspective: Prospective
Oversight: US Export: No

SUMMARY:
The body's immune system (fights infection) is known to decline during the aging process, resulting in an increased risk of catching infections. Vaccinations also are not as effective in protecting older people against infection as they are in younger people. The purpose of this study is to better understand how and why vaccines are not as effective in older people. The researchers believe that the immune response in older people who get a higher dose vaccine will be similar to the immune response in young adults who get the standard (lower) dose vaccine. This study is a substudy to a main study, evaluating flu vaccines in people 65 years and older. Volunteers who are in the main study will be asked if they will participate in the substudy. The substudy requires them to give 2 additional blood samples for an in-depth look at their immune response to the flu vaccine given in the main study. Substudy volunteers will have up to 3 clinic visits and participate up to 28 weeks.

DETAILED DESCRIPTION:
There is a need to increase protection against influenza conveyed to elderly persons by inactivated influenza virus vaccines. Serum antibody titer is the primary surrogate marker for immunity to influenza after vaccination; and increasing the antigen dose has been shown to increase the serum antibody response in vaccinated persons, including the elderly. However it is not known how the remainder of the immune system responds to the higher dose of influenza antigen. This study is linked to DMID protocols 04-100 and 05-0055. This study will be conducted as a substudy of DMID 04-100 at the University of Maryland, Baltimore. Subjects ages 65 years and older, who meet the entry criteria for the primary study, will be approached for participation in an immunology substudy of volunteers who receive a single intramuscular injection of either the high-dose or standard-dose of licensed 2004-2005 trivalent inactivated influenza vaccine. A minimum of 30 elderly subjects (with the possibility of up to 60 elderly subjects) will be enrolled for the substudy. The substudy will require an extra 100 ml (total blood draw of 120 ml) of blood drawn from the same 20 ml venipuncture obtained for hemagglutination inhibition assay (HAI) titers (as per the primary study) on days 0 and 28. To minimize adverse side effects, the additional 100 ml of blood required for the substudy will be obtained from the same venipuncture site from which the 20 ml blood will be obtained for HAI titers (i.e., if blood collection stops after the 20 ml for HAI are drawn, the researchers will not attempt to obtain additional blood from a separate venipuncture site). Subjects' blood will be evaluated for key humoral and cell-mediated immunity (CMI) responses to better understand the mechanisms underlying the predicted suboptimal immune responses to one or more of the three influenza vaccine antigens observed in the elderly. With regard to specific study objectives, blood samples will be submitted for the following analysis: (1) measurement of serum anti-HA (hemagglutinin) IgG and IgA antibodies by ELISA; (2) IgG antibody subclasses; (3) IgG and IgA avidity, (4) virus neutralizing functional assay; and (5) HAI antibody titer. Peripheral blood mononuclear cells (PBMC) isolated from these subjects will be evaluated for the following: (1) "central" and "effector" memory T cell responses, including their proliferative responses and cytokine production profiles by flow cytometry; (2) IFN-gamma production by ELISPOT, following specific antigenic stimulation; (3) measurement ex vivo of the frequency of circulating influenza-specific T cells by using commercially available MHC/tetramers and/or MHC/pentamers and flow cytometry; and (4) role of regulatory T cells in the modulation of influenza responses in the elderly. Studies for measurement ex vivo of the frequency of circulating influenza-specific T cells (by using commercially available MHC/tetramers and/or MHC/pentamers and flow cytometry) will concentrate on IFN-gamma, a cytokine shown by many investigators to play a central role in the host immune response to influenza antigens. If promising results are observed, other cytokines (e.g., IL-12, TNF-alpha) might also be evaluated in future investigations if sufficient cells and resources are available. Major factors involved in the decision to concentrate these studies on IFN-gamma include the need to remain focus in a defined set of scientific questions and the fact that we will only have access to a limited number of peripheral blood mononuclear cells (PBMCs) that might preclude the study of additional cytokines.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers who participate in Division of Microbiology and Infectious Diseases (DMID) study 04-100, "Comparisons of the Reactogenicity and Immunogenicity in Ambulatory Elderly Subjects of a Standard-Dose Fluzone® (15 µg HA/Virus Strain) and a High-Dose (60 µg HA/Virus Strain) of a Trivalent Inactivated Influenza Virus Vaccine" 2. Ambulatory medically stable persons at least 65 years of age on the date of vaccination 2. Provides written informed consent and will be available for all study visits 4. Able to understand and comply with planned study procedures Subjects will be considered ambulatory if they are not institutionalized, bedridden, or homebound. Medically stable subjects may have underlying illnesses such as hypertension, diabetes, ischemic heart disease, or hypothyroidism, but their symptoms/signs must be controlled with medical therapy. Subjects with acute febrile illnesses [oral temperature equal to or exceeding 99.5 degrees F (37.5 degrees C)] will be deferred until 3 days after illness resolution.

Exclusion Criteria:

1. Known allergy to eggs or other components of the vaccine (eg, thimerosal) 2. History of a severe reaction following influenza vaccination, systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to a vaccine containing the same substances 3. History of Guillain-Barré Syndrome 4. Immunosuppression as a result of underlying illness or treatment 5. Use of oral steroids, parenteral steroids, or high-dose inhaled steroids (> 800 µg per day of beclomethasone dipropionate or equivalent) within 1 month prior to vaccination 6. Use of other immunosuppressive or cytotoxic drugs or radiation therapy within the six months prior to vaccination 7. Active neoplastic disease or history of any hematologic malignancy in the past 5 years (except localized skin or prostate cancer that is stable in the absence of therapy) 8. Acute or chronic condition that (in the opinion of the Investigator) would render vaccination unsafe or would interfere with the evaluation of responses including, but not limited to the following: known chronic liver disease, significant renal disease, oxygen-dependent chronic lung disease, New York Heart Association Functional Class III or IV, unstable or progressive neurologic disorder, insulin-treated diabetes mellitus 9. Use of experimental vaccines or medications within the month prior to study entry, or expected use of experimental vaccines or medications during the entire study period, including the 6-month follow-up phone call, after inoculation with study vaccine 10. Use of experimental devices or participation in a medical procedure trial within the month prior to study entry, or expected use of experimental devices or participation in a medical procedure trial during the entire study period, including the 6-month follow-up phone call, after inoculation with study vaccine 11. Receipt of immunoglobulin or other blood product within 3 months prior to enrollment 12. Receipt of other licensed vaccines within the preceding 4 weeks or expected to receive a licensed vaccine within 1 month (prior to visit 2) following trial vaccination 13. Subject is enrolled in a conflicting clinical trial 14. Thrombocytopenia or bleeding disorder or therapy contraindicating intramuscular (IM) vaccination.

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-04-25 (Actual); Primary Completion 2005-05-30 (Actual); Study Completion 2005-05-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland School of Medicine - Center for Vaccine Development - Baltimore, Baltimore, Maryland, United States